CLINICAL TRIAL: NCT00158327
Title: The RELAX Trial: Reducing Limitations From Anxiety in Primary Care
Brief Title: Telephone-Based Care Management Program for Individuals With Anxiety Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Bruce Rollman, Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH059395 (NIH); R01MH059395 (NIH); RELAX; DSIR 82-SEPC
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Anxiety Disorders; Panic Disorder
Keywords: Primary Health Care
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): Participants will receive telephone-based collaborative care
  Interventions: Behavioral: Telephone-based collaborative care
- 2 (Active Comparator): Participants will receive usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Telephone-based collaborative care — Participants assigned to the telephone-based program will have a choice of what type of treatment they will receive. The choices will include pharmacotherapy, workbook training designed to help participants improve their coping skills, referral to a community mental health specialist, or some combination of these treatments. Participants will receive telephone calls one to two times every month for 12 months. During the calls, participants will be asked about their attitude toward and adherence to their treatment regimen. They will also be asked about recent episodes of anxiety they have experienced and what coping techniques they have used.
  Arms: 1
Behavioral: Usual care — Usual care may include one or more of several different treatments such as pharmacotherapy and cognitive behavioral therapy; the treatments will be chosen by participants' physicians and will be delivered for 12 months.
  Arms: 2

SUMMARY:
This study will determine the impact of a telephone-based care management program for primary care patients with panic disorder or generalized anxiety disorder.

DETAILED DESCRIPTION:
Numerous studies have shown that telephone-based collaborative care programs may be an effective way to monitor the quality of life of individuals with mental health issues such as anxiety disorders. With regular monitoring through telephone conversations, health care providers can gain information from their patients in a convenient forum. This study will determine whether a telephone-based care management program can improve anxiety symptoms, alcohol abuse, employment patterns, use of health care services, and health-related quality of life for individuals with panic disorder or generalized anxiety disorder (GAD).

Participants will be randomly assigned to receive either usual care or a telephone-based collaborative care program for 12 months. Usual care may include one or more of several different treatments such as pharmacotherapy and cognitive behavioral therapy; the treatments will be chosen by participants' physicians. Participants assigned to the telephone-based program will have a choice of what type of treatment they will receive; the choices will include pharmacotherapy, workbook training designed to help participants improve their coping skills, referral to a community mental health specialist, or some combination of these treatments.

Participants receiving usual care will continue their treatment for 12 months. After 12 months, these participants will undergo interviews and complete self-report scales for assessment of their anxiety symptoms, health care use, alcohol use, and quality of life. Their participation in the trial will end after 12 months.

Participants in the telephone intervention group will receive telephone calls 1 to 2 times every month for 12 months. During the calls, participants will be asked about their attitude toward and adherence to their treatment regimen. They will also be asked about recent episodes of anxiety they have experienced and what coping techniques they have used. Monthly follow-up calls will continue for an additional 12 months after the first year of the study; this will help determine the long-term effectiveness of the telephone-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of panic disorder or generalized anxiety disorder
* Score of 7 or higher on the Panic Disorder Severity Scale score OR a score of 14 or higher on the Structured Interview Guide for the Hamilton Anxiety Scale
* Life expectancy greater than 1 year
* Have a household telephone and can be contacted by phone for the duration of the study
* Able to read and write in English

Exclusion Criteria:

* Presently receiving treatment for a psychiatric disorder from a mental health specialist
* At risk for suicide
* History of bipolar disorder
* Dependence on alcohol or other substances within 6 months prior to study entry
* Organic anxiety syndromes, including those secondary to medical illness or drugs
* Unstable medical conditions that would interfere with the study
* Plan to leave their primary care source during the study or for 1 year after study completion

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2004-03; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (SF-36 MCS) | Measured at Month 12

SECONDARY OUTCOMES:
Generalized anxiety symptoms | Measured at Month 12
Panic disorder severity scale (PDSS) | Measured at Month 12
PHQ-9 | Measured at Month 12
Alcohol use | Measured at Month 12
Health services utilization | Measured at Month 12
Health care costs | Measured at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Bruce L. Rollman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Rollman BL, Herbeck Belnap B, Reynolds CF, Schulberg HC, Shear MK. A contemporary protocol to assist primary care physicians in the treatment of panic and generalized anxiety disorders. Gen Hosp Psychiatry. 2003 Mar-Apr;25(2):74-82. doi: 10.1016/s0163-8343(03)00004-5. PMID 12676419
- [Derived] Behringer T, Rollman BL, Herbeck-Belnap B, Houck PR, Mazumdar S, Schwarz EB. Impact of physician counseling and perception of teratogenic risks: a survey of 96 nonpregnant women with anxiety. Prim Care Companion CNS Disord. 2011;13(2):PCC.10m01028. doi: 10.4088/PCC.10m01028. PMID 21977355
- [Derived] Rollman BL, Fischer GS, Zhu F, Belnap BH. Comparison of electronic physician prompts versus waitroom case-finding on clinical trial enrollment. J Gen Intern Med. 2008 Apr;23(4):447-50. doi: 10.1007/s11606-007-0449-0. PMID 18373143